CLINICAL TRIAL: NCT06513962
Title: Triptorelin and Protection of Ovarian Reserve in Adolescents and Young Adults With Cancer
Brief Title: Triptorelin for the Prevention of Ovarian Damage in Adolescents and Young Adults With Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALTE2131; NCI-2024-05414 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE2131 (Other: Children's Oncology Group); COG-ALTE2131 (Other: DCP); ALTE2131 (Other: CTEP); UG1CA189955 (NIH)
Record Dates: First submitted 2024-07-03; First posted 2024-07-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (triptorelin) (Experimental): Patients receive triptorelin IM up to 14 days prior to standard chemotherapy. For patients whose chemotherapy exceeds 24 weeks, a second dose of triptorelin may be given 24 weeks after the first dose at the treating physician's discretion. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Survey Administration; Drug: Triptorelin Pamoate
- Arm B (usual care) (Active Comparator): Patients receive standard chemotherapy. Patients also undergo blood sample collection throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive standard chemotherapy
  Other Names: standard of care; standard therapy
  Arms: Arm B (usual care)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Other: Survey Administration — Ancillary studies
Drug: Triptorelin Pamoate — Given IM
  Other Names: Decapeptyl; Diphereline; Pamorelin; Trelstar; Triptorelin Embonate
  Arms: Arm A (triptorelin)

SUMMARY:
This phase III trial compares the effect of giving triptorelin vs no triptorelin in preventing ovarian damage in adolescents and young adults (AYAs) with cancer receiving chemotherapy with an alkylating agents. Alkylating agents are part of standard chemotherapy, but may cause damage to the ovaries. If the ovaries are not working well or completely shut down, then it will be difficult or impossible to get pregnant in the future. Triptorelin works by blocking certain hormones and causing the ovaries to slow down or pause normal activity. The triptorelin used in this study stays active in the body for 24 weeks or about 6 months after a dose is given. After triptorelin is cleared from the body, the ovaries resume normal activities. Adding triptorelin before the start of chemotherapy treatment may reduce the chances of damage to the ovaries.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of conducting a cross network, multi-site, randomized clinical trial of triptorelin among newly diagnosed adolescent and young adult (AYA) female cancer patients age < 40 years (exclusive of breast cancer).

II. Measure ovarian reserve via anti-Mullerian hormone (AMH) at 2-years post completion of alkylating agent-containing chemotherapy among randomized patients.

SECONDARY OBJECTIVES:

I. Collect information on the longitudinal trajectory of change in AMH and other ovarian hormone levels from cancer diagnosis to 2 years post cancer treatment completion among randomized patients.

II. Determine the feasibility of measuring estrogen deprivation symptoms (i.e., hot flashes, sexual dysfunction) menstrual pattern, and quality of life among randomized patients.

EXPLORATORY OBJECTIVE:

I. Establish a unique cohort of female AYA patients treated with alkylating agent chemotherapy and randomized to receive or not receive triptorelin, that can be followed long-term to study reproductive health concerns and outcomes as well as genetic risk factors for premature menopause.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive triptorelin intramuscularly (IM) up to 14 days prior to standard chemotherapy. For patients whose chemotherapy exceeds 24 weeks, a second dose of triptorelin may be given 24 weeks after the first dose at the treating physician's discretion. Patients also undergo blood sample collection throughout the study.

ARM B: Patients receive standard chemotherapy. Patients also undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* < 40 years of age at the time of enrollment
* Patient must be a post-menarchal female and report that their initial menstrual period occurred > 6 months prior to enrollment. (Current menstrual status is not part of the inclusion criteria.)
* Newly diagnosed with first cancer, exclusive of breast cancer.

  * Note: Apart from breast carcinoma, other tumor types originating in the breast are permitted (e.g., sarcoma, lymphoma).
* Planned treatment must include one or more of the following alkylating agents delivered with curative intent: cyclophosphamide, ifosfamide, procarbazine, chlorambucil, carmustine (BCNU), lomustine (CCNU), melphalan, thiotepa, busulfan, nitrogen mustard.
* For patients < 20 years of age at enrollment, the expected alkylator dose must be ≥ 4 g/m^2 cumulative cyclophosphamide equivalent dose (CED). For patients ≥ 20 years of age at enrollment, any planned alkylator dose is permitted. Eligible patients must receive at least one of the alkylators that contribute to CED.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Any planned radiation to the pelvis; or cranial radiation ≥ 30 gray (Gy) to the hypothalamus, inclusive of any total body irradiation (TBI).
* Planned bilateral oophorectomy. Note: A participant's desire to pursue alternative fertility preservation procedures (i.e., embryo, oocyte, or ovarian tissue cryopreservation) will be allowed (and in fact encouraged).
* Congenital syndromes associated with infertility and decreased ovarian reserve at baseline. For example: Turner's Syndrome, Fragile X premutation carriers, Down syndrome, etc.
* Pre-existing seizure disorder, congenital long QT syndrome, pseudotumor cerebri; history of pulmonary embolism, venous thrombosis, or myocardial infarction. Note: Contact study chairs if questions arise about other pre-existing conditions.
* Receipt of long acting (depot) GnRH agonists within 6 months before enrollment. In contrast, subcutaneous GnRH agonist used for oocyte retrieval is not an exclusion; oral and other hormonal contraceptive use is also not an exclusion. Note: Please see protocol for the concomitant therapy restrictions for patients during the study treatment period. See protocol for information about oral and other hormonal contractive use during the study treatment period.
* Prior receipt of systemic chemotherapy. However, steroids and intrathecal chemotherapy are permitted prior to study enrollment.
* Any prior radiation to the pelvis; or cranial radiation ≥ 30 Gy to the hypothalamus, inclusive of any total body irradiation (TBI).
* Patients who are pregnant are not eligible. A pregnancy test is required for female patients of childbearing potential.
* Lactating females who plan to breastfeed their infants for the duration of triptorelin therapy (24 weeks per dose).
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of triptorelin therapy (24 weeks per dose).

Max Age: 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of enrollments of newly diagnosed AYA female cancer patients age < 40 years | Up to 2 years post-chemotherapy
  Number of enrollments by the end of the DOD funded grant period, and ideally prior to Year 4 to enable greater duration of follow-up time. Will help determine if a larger efficacy study can be successfully completed as a cross network trial in a reasonable funding period.
Accrual rates of newly diagnosed AYA female cancer patients age < 40 years | Up to 2 years post-chemotherapy
  Accrual rates of newly diagnosed AYA female cancer patients age < 40 years. Over the second half of the funding period, demonstrate a positive trajectory in accrual rates that provides data to inform future funding proposals that would seek to complete the overall larger study within a typical 5-year funding period.
Anti-mullerian hormone (AMH) levels | At 2 years post-chemotherapy
  AMH values will be examined to confirm that the combined variability of AMH in both arms is consistent with our a priori assumptions.

SECONDARY OUTCOMES:
Longitudinal AMH along with other ovarian hormone levels | Up to 2 years post-chemotherapy
  These measurements will help inform rates of missingness. Will be used to estimate the longitudinal trajectory of change in these hormones by triptorelin randomization status.
Estrogen deprivation symptoms: Hot flashes | Up to 2 years post-chemotherapy
  Estrogen deprivation symptoms include hot flashes. The Patient-Reported Outcomes version of the Common Terminology for Adverse Events (PRO-CTCAE) will be used to collect information on the frequency and interference of hot flashes.
Estrogen deprivation symptoms: Headaches | Up to 2 years post-chemotherapy
  Estrogen deprivation symptoms include headaches. The Patient-Reported Outcomes version of the Common Terminology for Adverse Events (PRO-CTCAE) will be used to collect information on the frequency and interference of headaches.
Estrogen deprivation symptoms: Vaginal/vulvar symptoms | Up to 2 years post-chemotherapy
  Estrogen deprivation symptoms include vaginal/vulvar symptoms. The Patient-Reported Outcomes version of the Common Terminology for Adverse Events (PRO-CTCAE) will be used to collect information on the frequency and interference of vaginal/vulvar symptoms. The PROMIS Sexual Function and Satisfaction version (v) 2.0 Brief Profile - Female (PROMIS SexFS) will be used to evaluate vaginal and vulvar discomfort, pain, and lubrication.
Estrogen deprivation symptoms: Sexual function | Up to 2 years post-chemotherapy
  Estrogen deprivation symptoms include sexual function. The Patient-Reported Outcomes version of the Common Terminology for Adverse Events (PRO-CTCAE) will be used to collect information on the frequency and interference of sexual function. The PROMIS Sexual Function and Satisfaction version (v) 2.0 Brief Profile - Female (PROMIS SexFS) will be used to evaluate sexual activity, desire, and satisfaction among all participants.
Sexual Health | Up to 2 years post-chemotherapy
  Sexual dysfunction will be assessed using PROMIS SexFS.
Menstrual patterns | Up to 2 years post-chemotherapy
  Menstrual patterns will be assessed using standard items and characterized according to the Staging of Reproductive Aging Workshop criteria.
Global health-related quality of life: Anxiety | Up to 2 years post-chemotherapy
  Global health-related quality of life will be assessed using the PROMIS 29 Profile v2.1, which includes assessment of anxiety. For adolescent participants, the PROMIS Pediatric Profile-25 v2.0 will be used to measure health domains.
Global health-related quality of life: Fatigue | Up to 2 years post-chemotherapy
  Global health-related quality of life will be assessed using the PROMIS 29 Profile v2.1, which includes assessment of fatigue. For adolescent participants, the PROMIS Pediatric Profile-25 v2.0 will be used to measure health domains.
Global health-related quality of life: Depression | Up to 2 years post-chemotherapy
  Global health-related quality of life will be assessed using the PROMIS 29 Profile v2.1, which includes assessment of depression. For adolescent participants, the PROMIS Pediatric Profile-25 v2.0 will be used to measure health domains.
Global health-related quality of life: Sleep disturbance | Up to 2 years post-chemotherapy
  Global health-related quality of life will be assessed using the PROMIS 29 Profile v2.1, which includes assessment of sleep disturbance. For adolescent participants, the PROMIS Pediatric Profile-25 v2.0 will be used to measure health domains, with the addition of the PROMIS Pediatric Sleep Disturbance 4a scale.
Global health-related quality of life: Participation in social activities | Up to 2 years post-chemotherapy
  Global health-related quality of life will be assessed using the PROMIS 29 Profile v2.1, which includes assessment of participation in social activities. For adolescent participants, the PROMIS Pediatric Profile-25 v2.0 will be used to measure health domains.

OTHER OUTCOMES:
Reproductive concerns | Up to 2 years post-chemotherapy
  The reproductive concerns after cancer scale will be used for fertility potential and acceptance.
Reproductive outcomes | Up to 2 years post-chemotherapy
  Reproductive outcomes will be assessed using selected questions from the US Centers for Disease Control and Prevention's National Health and Nutrition Examination Survey's (NHANES) Reproductive Health module.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Chow, Principal Investigator — Children's Oncology Group
Locations (176):
- United States (175):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Healthcare Mission Cancer and Blood - Pella, Pella, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
- CancerCare Manitoba, Winnipeg, Manitoba, Canada